CLINICAL TRIAL: NCT04229966
Title: A Real World, Multicenter, Prospective, Observational Study to Compare Effectiveness of Surgical Treatments in Patients With Acute Epidural Hematoma
Brief Title: Prospective, Observational Real-world Treatments of AEDH in Large-scale Surgical Cases
Acronym: PORTALS-AEDH
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Clinical Research Institute, Shanghai Jiao Tong University School of Medicine (Unknown); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PORTALS-AEDH
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Epidural Hematoma; Decompressive Craniectomy; Craniotomy
MeSH Terms: conditions — Hematoma, Epidural, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, prospective, and observational real-world study aimed at investigating the current situation of surgical treatments and prognosis for acute epidural hematoma in China, and analyzing the optimization of therapy.

DETAILED DESCRIPTION:
The incidence of Acute Epidural Hematoma (AEDH) among traumatic brain injury (TBI) patients has been reported to be in the range of 2.7 to 4%. The mortality in patients in all age groups and GCS scores undergoing surgery for evacuation of EDH is approximately 10%.

Most people with EDH are generally expected to have a good clinical outcome with the prompt and correct treatment. However, AEDH still represents a potentially life-threatening condition when a local mass effect exists due to rapidly elevated intracranial pressure (ICP) resulted from the rapid build-up of blood. Brain hernia and cerebral infarction might occur and lead to a terrible clinical outcome. In addition, there is a set of patients who experience clinical deterioration after an initial hematoma-evacuation craniotomy because of secondary brain injuries, including massive cerebral infarction (MCI), additional decompressive craniectomy is recommended as soon as possible.

Although DC can reduce the morbidity and mortality in critically ill patients with a sTBI, the removal of the bone flap is not necessary for the majority of patients with AEDH, because of the relatively low incidence of MCI secondary to AEDH. Recommendations indicated an epidural hematoma greater than 30 ml should be surgically evacuated regardless of the patient's GCS score. Although craniotomy provides a complete evacuation to remove the clot of the hematoma, there are insufficient data to support a specific surgical treatment method. The choice of operative technique is influenced by the surgeon's expertise, training, and evaluation of a particular situation. Therefore, there is a clinical rationale for investigating the current status of surgical treatments and prognosis for AEDH, thereby providing a reliable reference for the optimization of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Clear medical history of traumatic brain injury;
2. within 12 hours after injury;
3. Supratentorial unilateral acute epidural hematoma on first head CT scan examination;
4. The admitting neurosurgeon considers that the epidural hematoma needs to be evacuated with surgical treatment;
5. With informed consent to surgery and trial participation.

Exclusion Criteria:

1. Previous intracranial surgery prior to trauma;
2. Patients with a score of 3 on the GCS, with bilateral fixed and dilated pupils, bleeding diathesis or defective coagulation, or an injury that was deemed to be unsurvivable;
3. CT demonstrates associated other intracranial hematomas e.g. subdural, intracerebral hemorrhage, or large size infarction, which are the main causes of operation;
4. Patients who had injury of the oculomotor nerve;
5. Severe pre-existing disability or severe co-morbidity which would lead to a poor outcome even if the patient is supposed to a good recovery from the TBI;
6. Pregnant female.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population who were diagnosed with acute epidural hematoma and necessary for undergoing evacuation of an acute epidural hematoma.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
GOSE (extended Glasgow Outcome Scale) scores | at 6 months post-injury
  The primary outcome is indicated by the long-term functional outcomes, including overall mortality and the score on the Extended Glasgow Outcome Scale (GOS-E), "Extended Glasgow Outcome Scale" is the unabbreviated scale title. The minimum value of scale is score 1, and maximum value is scored 8, higher scores mean a better outcome and lower scores mean worse outcome. Specific scored as follows:
  1. death;
  2. persistent vegetative state;
  3. lower severe disability;
  4. upper severe disability; (stratum 3 and 4 were considered as severe disability, with permanent requirement for help with daily living);
  5. lower moderate disability;
  6. upper moderate disability; (stratum 5 and 6 were considered as mild disability, without a need for assistance in everyday life, that might, however, require special equipment for employment);
  7. lower good recovery;
  8. upper good recovery (stratum 7 and 8 were considered as good recovery).

SECONDARY OUTCOMES:
incidence of post-operative cerebral infarction | within 6 months post-injury
  The incidence of traumatic AEDH post-operative cerebral infarction within 6 months post-injury, which is primarily diagnosed by independent radiologists with CT or MRI examination.
incidence of additional craniocerebral surgery | within 6 months post-injury
  The incidence of additional craniocerebral surgery within 6 months post-injury, related to clinical deterioration after initial surgical treatment of AEDH.
length of stay in ICU and hospital | within 6 months post-injury
  The duration of hospitalization after initial surgery within 6 months post-injury, including ICU and hospital stays.
detailed economic evaluation | within 6 months post-injury
  Total medical expense related to treatment of AEDH, including the costs of operations, hospitalization and rehabilitation within 6 months post-injury.
incidence of serious adverse events | within 6 months post-injury
  Serious adverse events (SAE) is defined as an untoward occurrence that:
  1. results in death
  2. is life-threatening
  3. requires hospitalisation or prolongation of existing hospitalization
  4. results in persistent or significant disability or incapacity
  5. is otherwise considered medically significant by the investigator.
quality of life (EQ-5D-5L) | at 6 months post-injury
  Unabbreviated scale title is "5-level EuroQol five dimensions" questionnaire. The EQ-5D is a generic instrument for describing and valuing health. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
MMSE (mini-mental state examination) scores | at 6 months post-injury
  MMSE (mini-mental state examination) scores at 6 months post-injury.

CONTACTS AND LOCATIONS:
Overall Officials: Jiyao Jiang, Professor, Study Chair — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Department of Neurosurgery, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Bullock MR, Chesnut R, Ghajar J, Gordon D, Hartl R, Newell DW, Servadei F, Walters BC, Wilberger JE; Surgical Management of Traumatic Brain Injury Author Group. Surgical management of acute epidural hematomas. Neurosurgery. 2006 Mar;58(3 Suppl):S7-15; discussion Si-iv. PMID 16710967
- [Background] Li LM, Kolias AG, Guilfoyle MR, Timofeev I, Corteen EA, Pickard JD, Menon DK, Kirkpatrick PJ, Hutchinson PJ. Outcome following evacuation of acute subdural haematomas: a comparison of craniotomy with decompressive craniectomy. Acta Neurochir (Wien). 2012 Sep;154(9):1555-61. doi: 10.1007/s00701-012-1428-8. Epub 2012 Jun 30. PMID 22752713
- [Background] Lin H, Wang WH, Hu LS, Li J, Luo F, Lin JM, Huang W, Zhang MS, Zhang Y, Hu K, Zheng JX. Novel Clinical Scale for Evaluating Pre-Operative Risk of Cerebral Herniation from Traumatic Epidural Hematoma. J Neurotrauma. 2016 Jun 1;33(11):1023-33. doi: 10.1089/neu.2014.3656. Epub 2016 Jan 28. PMID 25393339
- [Background] Wang WH, Hu LS, Lin H, Li J, Luo F, Huang W, Lin JM, Cai GP, Liu CC. Risk factors for post-traumatic massive cerebral infarction secondary to space-occupying epidural hematoma. J Neurotrauma. 2014 Aug 15;31(16):1444-50. doi: 10.1089/neu.2013.3142. Epub 2014 Jun 25. PMID 24773559
- [Derived] Yang C, Hui J, Xie L, Feng J, Jiang J. Comparative effectiveness of different surgical procedures for traumatic acute epidural haematoma: study protocol for Prospective, Observational Real-world Treatments of AEDH in Large-scale Surgical Cases (PORTALS-AEDH). BMJ Open. 2022 Mar 9;12(3):e051247. doi: 10.1136/bmjopen-2021-051247. PMID 35264341